CLINICAL TRIAL: NCT06424288
Title: EASi-HF Preserved - A Phase III Double-blind, Randomised, Parallel-group Superiority Trial to Evaluate Efficacy and Safety of the Combined Use of Oral Vicadrostat (BI 690517) and Empagliflozin Compared With Placebo and Empagliflozin in Participants With Symptomatic Heart Failure (HF: NYHA II-IV) and Left Ventricular Ejection Fraction (LVEF) ≥40%
Brief Title: A Study to Test Whether Vicadrostat in Combination With Empagliflozin Helps People With Heart Failure
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1378-0020; 2023-509706-30-00 (Registry Identifier: CTIS); U1111-1302-4422 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-05-10; First posted 2024-05-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- vicadrostat/empagliflozin (Experimental)
  Interventions: Drug: vicadrostat; Drug: empagliflozin
- placebo/empagliflozin (Placebo Comparator)
  Interventions: Drug: empagliflozin; Drug: placebo

INTERVENTIONS:
Drug: vicadrostat — vicadrostat
  Arms: vicadrostat/empagliflozin
Drug: empagliflozin — empagliflozin
Drug: placebo — placebo matching vicadrostat
  Arms: placebo/empagliflozin

SUMMARY:
This study is open to adults aged 18 or above legal age with heart failure. People can join the study if they have heart failure symptoms and a left ventricular ejection fraction (LVEF) of 40% or more. The purpose of this study is to find out whether vicadrostat (BI 690517) in combination with empagliflozin helps people with heart failure.

Participants are put into 2 groups by chance. Every participant has an equal chance of being in each group. The groups are:

* Vicadrostat/empagliflozin group: participants take vicadrostat/empagliflozin as tablets once a day.
* Placebo/empagliflozin group: participants take placebo/empagliflozin as tablets once a day.

Participants can stay in the study as long as they benefit from treatment and can tolerate it. During this time, they visit their doctors regularly. The doctors regularly check participants' health and take note of any unwanted effects. The study staff may also contact the participants by phone. Participants also regularly answer questions about their well-being.

The study does not have a fixed duration. It continues until there is enough data to see if the treatment is working.

ELIGIBILITY:
Inclusion criteria:

1. At least 18 years old and at least of the legal age of consent in countries where it is greater than 18 years
2. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
3. Male or female participants. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per International Conference on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria and instructions on the duration of their use is provided in the participant information
4. Chronic Heart failure (HF) diagnosed at least 3 months before Visit 1, and in New York Heart Association (NYHA) class II-IV at Visit 1, with left ventricular ejection fraction (LVEF) ≥40% per local reading. A historical LVEF may be used if it was measured within 12 months prior to Visit 1, or the LVEF may be measured after study consent has been obtained and before randomisation at Visit 2
5. Presence of structural heart abnormality (confirmed by any imaging modality; i.e. echocardiography at Visit 1, as defined by left ventricular hypertrophy or left atrial enlargement). Historical imaging may be used if performed within 12 months prior to Visit 1, or imaging may be completed after study consent has been obtained and before Visit 2
6. Elevated N-terminal pro-brain natriuretic peptide (NT-proBNP) at Visit 1, analysed at the central laboratory at Visit 1:

   1. in participants with body mass index (BMI) <27 kg/m²: ≥300 pg/mL for participants without atrial fibrillation (Afib) or atrial flutter (Aflutter) (at Visit 1 electrocardiogram (ECG)) and ≥900 pg/mL for participants with Afib or Aflutter (at Visit 1 ECG)
   2. in participants with BMI ≥27 kg/m² to <35 kg/m²: ≥220 pg/mL for participants without Afib or Aflutter (at Visit 1 ECG) and ≥660 pg/mL for participants with Afib or Aflutter (at Visit 1 ECG)
   3. in participants with BMI ≥35 kg/m²: ≥125 pg/mL for participants without Afib or Aflutter (at Visit 1 ECG) and ≥375 pg/mL for participants with Afib or Aflutter (at Visit 1 ECG)
7. At least one of the following:

   * Currently treated with diuretic therapy e.g. loop diuretics or thiazides, and on a stable dose for at least 1 week prior to Visit 1
   * Documented hospitalisation for HF within 6 months prior to Visit 1
   * Elevated NT-proBNP at Visit 1, analysed at the central laboratory at Visit 1

     * in participants without Afib or Aflutter (at Visit 1 ECG): ≥900 pg/mL
     * for participants with Afib or Aflutter (at Visit 1 ECG): ≥1800 pg/mL
   * Urine albumin-to-creatinine ratio (UACR) ≥30 mg/g, analysed at the central laboratory at Visit 1
8. Treated according to best possible standard of care (SOC) (disregarding Sodium-dependent glucose co-transporter 2 inhibitors (SGLT2is) and Mineralocorticoid receptor antagonists (MRAs)) in accordance with applicable HF local/international guidelines and judgment of the investigator Further inclusion criteria apply.

Exclusion criteria:

1. Treatment with an mineralocorticoid receptor antagonist (MRA) (e.g. spironolactone, eplerenone, finerenone) within 14 days prior to Visit 1 or requiring such treatment before randomisation or planned during the trial based on the judgment of the investigator. Treatment with MRA should not be interrupted with the intention of enrolment into the study
2. Treatment with amiloride, or other potassium-sparing diuretic within 14 days prior to Visit 1 or requiring such treatment before randomisation or planned during the trial based on the judgment of the investigator
3. Receiving the following treatments:

   * a direct renin inhibitor (e.g. aliskiren) at Visit 2
   * more than one angiotensin-converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB) or angiotensin receptor-neprilysin inhibitor (ARNI) used simultaneously at Visit 2
   * In case of acute decompensated HF:

     * i.v. inotrope, i.v. vasodilating drug (e.g. nitrate, nitroprusside), or i.v. natriuretic peptide (e.g. nesiritide, carperitide), or mechanical support (e.g. intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, any ventricular assist device) within 24 hours prior to randomisation (Visit 2)
     * i.v. diuretic with a dose that has been increased/intensified within 6 hours prior to randomisation (a stable dose of an i.v. diuretic is not exclusionary)
   * Systemic mineralocorticoid replacement therapy (e.g. fludrocortisone) at Visit 2
   * Other aldosterone synthase inhibitors, e.g. baxdrostat at Visit 2 or planned during the trial
4. Myocardial infarction (MI), transient ischemic attack (TIA), stroke, coronary artery bypass graft (CABG) surgery, heart valve surgery/intervention or any other major surgery (major according to the investigator's assessment) within 90 days prior to Visit 2, or scheduled for major elective surgery (e.g. hip replacement, coronary artery bypass graft surgery/CABG)
5. Percutaneous coronary intervention (PCI) ( scheduled or unscheduled) or any angiography using iodinated contrast agents in the 7 days prior to Visit 2
6. Heart transplant recipient, awaiting heart transplant, or currently implanted left ventricular assist device (LVAD)
7. Known cardiomyopathy based on infiltrative diseases (e.g. amyloidosis), accumulation diseases (e.g. haemochromatosis, Fabry disease), muscular dystrophies, hypertrophic obstructive cardiomyopathy or genetic hypertrophic cardiomyopathy,known pericardial constriction, or cardiomyopathy with potentially reversible cause such as stress or peripartum cardiomyopathy or cardiomyopathy induced by chemotherapy within the 12 months prior to Visit 1 and until Visit 2
8. Acute inflammatory heart disease, such as acute myocarditis, within the 90 days preceding prior to Visit 1 and until Visit 2
9. Known severe valvular heart disease (obstructive or regurgitant), as per investigator's judgment, or valvular heart disease scheduled for surgical or invasive procedures at Visit 1, or anticipated invasive treatment during the study Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2028-05-22 (Estimated); Study Completion 2028-05-22 (Estimated)

PRIMARY OUTCOMES:
Time to first event of Cardiovascular (CV) death, hospitalisation for heart failure (HHF) or urgent heart failure (HF) visit | up to 42 months

SECONDARY OUTCOMES:
Key secondary endpoint: Time to first event of CV death or HHF | up to 42 months
Key secondary endpoint: Occurrence of HHFs (first and recurrent) | up to 42 months
Key secondary endpoint: Absolute change from baseline in Kansas City Cardiomyopathy Questionnaire Total Symptom Score (KCCQ-TSS) at Week 32 | at baseline, at week 32
  The Kansas City Cardiomyopathy Questionnaire is a patient-reported outcome instrument for use in clinical investigations in heart failure.
  The Total Symptom Score measures the following aspects of symptom experience in two domain scores:
  The "Symptom Frequency Domain" assesses frequency of the following experiences:
  * Lower extremity swelling in the morning
  * Fatigue limiting patients' ability to do what they want
  * Dyspnea limiting patients' ability to do what they want
  * Dyspnea forcing patients to sleep upright/elevated
  The "Symptom Burden Domain" assesses bothersomeness of the following symptoms:
  * Fatigue
  * Dyspnea
  * Lower extremity swelling All KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Key secondary endpoint: Time to CV death | up to 42 months
Key secondary endpoint: Time to all-cause mortality | up to 42 months
Time to first HHF | up to 42 months
Time to first occurrence of death from kidney failure, chronic dialysis* or renal transplant or onset of sustained reduction of ≥50% eGFR from baseline** or onset of sustained eGFR (CKD-EPI)cr <10 mL/min/1.73 m2 (composite renal endpoint) | up to 42 months
  * chronic dialysis is defined as dialysis continuing for at least 30 days
  ** using the Chronic Kidney Disease Epidemiology Collaboration creatinine equation ((CKD-EPI)cr)
Absolute change from baseline in KCCQ Clinical Summary Score (KCCQ-CSS) at Week 32 | at baseline, at week 32
  The KCCQ Clinical Summary Score is a composite of the Total Symptom Score and Physical Limitations Score.
  The "Physical Limitations Score" measures the following physical limitations:
  * Dressing
  * Showering/bathing
  * Walking one block on level ground
  * Doing yardwork, housework or carrying groceries
  * Climbing a flight of stairs without stopping
  * Hurrying or jogging as if to catch a bus All KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Absolute change from baseline in KCCQ-TSS at Week 52 | at baseline, at week 52
Absolute change from baseline in KCCQ-OSS at Week 32 | at baseline, at week 32
  The Kansas City Cardiomyopathy Questionnaire - overall summary score (KCCQ-OSS) is a combination of the symptom [domain], physical limitations, social limitations, and quality of life domains.
  All KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Absolute change from baseline in KCCQ-OSS at Week 52 | at baseline, at week 52
Absolute change from baseline in systolic blood pressure (SBP) [mmHg] at Week 32 in participants with baseline SBP ≥130 mmHg | at baseline, at week 32
Absolute chance from baseline in diastolic blood pressure (DBP) [mmHg] at Week 32 in participants with baseline DBP ≥80 mmHg | at baseline, at week 32

CONTACTS AND LOCATIONS:
Locations (626):
- United States (93):
  - Diagnostic and Medical Clinic, Mobile, Alabama
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - Velocity Clinical Research-Chula Vista, Chula Vista, California
  - University of California Irvine, Orange, California
  - North America Research Institute, San Dimas, California
  - Orange County Research Center, Tustin, California
  - Amicis Research Center (ARC), Valencia, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Bay Area Cardiology, Brandon, Florida
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - Cardiology Associates Research Co., Daytona Beach, Florida
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Velocity Clinical Research-Hallandale Beach-67888, Hallandale, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - East Coast Institute for Research, LLC - Jacksonville, Jacksonville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Clearwater Cardiovascular Consultants-Largo-69917, Largo, Florida
  - University of Miami, Miami, Florida
  - Sacred Heart Medical Specialty Group, Miramar Beach, Florida
  - Advanced Research for Health Improvement, LLC, Naples, Florida
  - Southwest Florida Research, LLC, Naples, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Ocala Research Institute, Inc, Ocala, Florida
  - Charlotte Cardiovascular Institute, PA, Port Charlotte, Florida
  - East Coast Institute for Research, LLC-Saint Augustine-63032, Saint Augustine, Florida
  - University of South Florida, Tampa, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Cozy Research LLC, Wesley Chapel, Florida
  - Clinical Site Partners, LLC, Winter Park, Florida
  - Atlanta Clinical Research Centers, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - NSC Research Inc, Johns Creek, Georgia
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Illinois Masonic Hospital, Chicago, Illinois
  - Chicago Medical Research, Hazel Crest, Illinois
  - Clinical Investigation Specialists, Inc.-Libertyville-69941, Libertyville, Illinois
  - AMR Park Ridge, Park Ridge, Illinois
  - Midwest Cardiovascular Research and Education Foundation, Elkhart, Indiana
  - St. Francis Medical Group-Indiana Heart Physicians, Inc, Indianapolis, Indiana
  - Indiana Medical Research Institute, Merrillville, Indiana
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - Reid Hospital, Richmond, Indiana
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - West Houston Area Clinical Trial Consultants, LLC, Wichita, Kansas
  - Norton Heart Specialists, Louisville, Kentucky
  - Grace Research, LLC-Bossier City-51040, Bossier City, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Grace Research, LLC-Shreveport-64616, Shreveport, Louisiana
  - Louisiana Heart Center - Slidell, Slidell, Louisiana
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - AMR Dearborn, Dearborn, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Trinity Health Michigan D/B/A Michigan Heart, Ypsilanti, Michigan
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - Jackson Heart Clinic, P.A., Jackson, Mississippi
  - Kansas City VA Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - St. Louis Heart and Vascular, P.C., St Louis, Missouri
  - Velocity Clinical Research-Lincoln-69943, Lincoln, Nebraska
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - Garden State Heart Care, PC, Manalapan, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - NYU Langone Health, New York, New York
  - Mount Sinai Hospital-New York-52529, New York, New York
  - Cardiac Care and Vascular Medicine, PLLC, The Bronx, New York
  - Medication Management, LLC, Greensboro, North Carolina
  - WakeMed, Raleigh, North Carolina
  - K and R Research LLC, Marion, Ohio
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - Bon Secours Medical Group Greenville Specialty Care, LLC, Greenville, South Carolina
  - Monument Health, Rapid City, South Dakota
  - Helios CR Inc, Jackson, Tennessee
  - East Coast Institute For Research LLC, Jefferson City, Tennessee
  - Pharmatex Research, Amarillo, Texas
  - Amarillo Heart Clinical Research Institute, Incorporated, Amarillo, Texas
  - Texas Health Research and Education Institute, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Helios CR Inc, Fort Worth, Texas
  - Private Practice Leadership, LLC, Katy, Texas
  - Texas Cardiology Research Center PLLC, Kingwood, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - North Texas Research Associates, McKinney, Texas
  - Texas Institute Of Cardiology, McKinney, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Carient Heart and Vascular, Manassas, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Selma Medical Associates, Winchester, Winchester, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Drug Research and Analysis Corporation, Madison, Wisconsin
  - ProHealth Care Research Institute and Cardiology Associates, Waukesha, Wisconsin
- Argentina (32):
  - Inst de Inv Clinicas-Bahia Blanca, Bahía Blanca
  - Swiss Medical Center Barrio Parque, Buenos Aire
  - Centro de Investigaciones Metabolicas (CINME)-Ciudad Autonoma Buenos Aires-41221, Ciudad Autonoma Buenos Aires
  - Mautalen- Salud e Investigacion, Ciudad Autonoma Buenos Aires
  - Centro Medico Dra Laura Maffei, Ciudad Autonoma Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma Buenos Aires
  - Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Glenny Corp. S.A. Bioclinica Argentina, Ciudad Autonoma Buenos Aires
  - Centro Medico Viamonte, Ciudad Autonoma de Bs As
  - Hospital Italiano de Buenos Aires, Ciudad Autónoma de Bs As
  - Instituto Medico Elsa Perez SRL (IMEP), Ciudadela
  - Clinica Coronel Suárez, Coronel Suárez
  - Sanatorio Allende S.A., Córdoba
  - Sanatorio Privado Duarte Quiros De Clinica Colombo SA, Córdoba
  - Well Medica, Córdoba
  - Instituto Médico DAMIC S.R.L., Córdoba
  - Centro Medico Luquez, Córdoba
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata
  - Hospital Universitario Austral, Pilar
  - Instituto de Investigaciones Clínicas de Quilmes, Quilmes
  - DIM Clinica Privada, Ramos Mejía
  - Instituto de Investigaciones Clinicas de Rosario, Rosario
  - Instituto CAICI, Rosario
  - Centro Cardiovascular Salta, Salta
  - Corporacion Medica de Gral. San Martin S.A., San Martín
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
  - Centro Modelo de Cardiologia, San Miguel de Tucumán
  - Clinica Mayo, San Miguel de Tucumán
  - Instituto de Investigaciones Clinicas San Nicolas, San Nicolás
  - Centro de Investigaciones Clínicas del Litoral, Santa Fe
  - CEMEDIC - Centro de Especialidades Medicas, Villa Luro
- Australia (13):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Pendlebury Research, Kotara, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Prince Charles Hospital, Chermside, Queensland
  - John Flynn Private Hospital, Tugun, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Total Cardiovascular Care, Frankston, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Mount Hospital, Perth, Western Australia
- Belgium (6):
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Sint-Lucas, Ghent
  - Grand Hôpital de Charleroi, Gilly
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
- Brazil (38):
  - Centro de Pesquisa Clínica do Coração, Aracaju
  - Hospital Felicio Rocho, Belo Horizonte
  - Hospital Vera Cruz, Belo Horizonte
  - Cardresearch Cardiologia Assistencial e de Pesquisas Ltda, Belo Horizonte
  - Hospital Universitário São Francisco na Providência de Deus, Bragança Paulista
  - L2IP -Instituto de Pesquisas Clínicas Ltda., Brasília
  - Hospital DF Star, Brasília
  - Hospital do Coracao do Brasil, Brasília
  - CECAP - Centro de Cardiologia Clínica, Brasília
  - Hospital Brasilia, Brasília
  - Hospital Angelina Caron, Campina Grande do Sul
  - IPECC - Instituto de Pesquisa Clínica de Campinas, Campinas
  - Centro Especializado em Cardiol Loema Instituto de Pesq Clin, Campinas
  - Hospital do Rocio, Campo Largo
  - PUC Trials - Núcleo de Pesquisa Clínica da Escola de Medicina da PUC-PR, Curitiba
  - Via Medica, Goiânia
  - ICM - Instituto do Coracao de Marilia, Marília
  - Instituto Atena de Pesquisa Clinica, Natal
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Universidade Federal do Rio Grande do Sul, Porto Alegre
  - Hospital Mae de Deus, Porto Alegre
  - Hospital Esperança Recife, Recife
  - Clinicor Clínica Cardiológica LTDA/ Cardio Prime - CAPED, Ribeirão Preto
  - Hospital das Clínicas FMRP-USP, Ribeirão Preto
  - Instituto Brasil de Pesquisa Clinica (IBPClin), Rio de Janeiro
  - Ruschel Medicina e Pesquisa Clínica, Rio Do Janeiro
  - Hospital Cardio Pulmonar, Salvador
  - Pesquisare, Santo André
  - Praxis Pesquisa Medica, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, Sao Jose Rio Preto
  - Hospital Sao Domingos, São Luís
  - Centro de Pesquisa Clinica - CPCLIN, São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica, São Paulo
  - Eurolatino Pesquisas Médicas Ltda., Uberlândia
  - CEDOES - Diagnóstico e Pesquisa,Vitória, Vitória
  - Integral Pesquisa e Ensino, Votuporanga
- Bulgaria (30):
  - Medical Center Doktor Staykov Ltd., Burgas
  - Diamedical Medical Center 2013, Dimitrovgrad
  - MHAT Ivan Skenderov EOOD, Gotse Delchev
  - Medical Center Rodopimed EOOD, Kardzhali
  - Medical Center Hera - Kyustendil EOOD, Kyustendil
  - Ambulatory Individual Practice for Cardiology Specialized Medical Care, Pernik
  - Medical Center Medconsult Pleven OOD, Pleven
  - MHAT Heart and brain, Pleven
  - Ambulatory for Individual Practice for Specialized Medical Care in Cardiology - Dr Nikolay Iliev, Pleven
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - Medical Center Rusemed EOOD, Rousse
  - National Multiprofile Transport Hospital "Tzar Boris III", Sofia
  - Medical Center For Specialized Medical Help In Cardiovascular Diseases OOD, Sofia
  - Alexandrovska University Hospital, Sofia
  - Diagnostic Consultative Center Alexandrovska, Sofia
  - University Multidisciplinary Hospital for Active Treatment Sveta Ekaterina EAD, Sofia
  - Medical Center Hera EOOD, Sofia
  - UMHAT "Tsaritsa Yoanna-ISUL" EAD, Sofia
  - ASOMHIDC - Individual practice "Cardio Tonus" EOOD, Sofia
  - Multiprofile Hospital MHATEM 'Pirogov', Sofia, Sofia
  - Diagnostic Consultation Center XX-Sofia EOOD, Sofia
  - MHAT "St. Sofia", Sofia
  - Kalimat Medical Center Ltd., Sofia
  - Medical Center Intermedica Ltd., Sofia
  - Medical Center Medicabilis Ltd., Sofia
  - UMHAT Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
  - Medical Center Zara-Med EOOD, Stara Zagora
  - Diagnostichno-Consultativen Center Chaika EOOD, Varna
  - Medical Centre Nevromedics EOOD, Veliko Tarnovo
  - MHAT St Panteleimon, Yambol
- Canada (18):
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Curnew Medicine Professional Corporation, Hamilton, Ontario
  - KMH Cardiology Centres (Mississauga), Mississauga, Ontario
  - Oakville Trafalgar Memorial Hospital, Oakville, Ontario
  - James Cha, MD, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - CardioQuest Research Centre, Sarnia, Ontario
  - KMH Cardiology Centers (Hamilton), Stoney Creek, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - ViaCar Recherches Cliniques Inc. (Greenfield Park), Greenfield Park, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Diex Recherche (Trois-Rivieres), Trois-Rivières, Quebec
  - Royal Alexandra Hospital, Edmonton
  - Health Sciences North, Greater Sudbury
  - Clinical Research Solutions Inc. (Kitchener), Kitchener
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal
  - Montreal General Hospital - McGill University Health Centre, Montreal
  - CardioVasc HR Inc., Saint-Jean-sur-Richelieu
- Chile (5):
  - Quantum Research Santiago, Puerto Varas, Puerto Varas
  - Sociedad Medica Cardiologica El Llano, Santiago
  - Hospital Las Higueras, Talcahuano
  - CECMI Ltda, Temuco
  - CINVEC - Centro de Investigacion Clinica V Reg.,Vina del Mar, Viña del Mar
- China (75):
  - The First Affiliated Hospital of Baotou Medical College, Baotou
  - Baotou Central Hospital, Baotou
  - Beijing AnZhen Hospital, Capital Medical University, Beijing
  - Cardiovascular Institute and Fu Wai Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Jilin Province People's Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - China-Japan Union Hospital of Jilin University, Changchun
  - Changde Second People's Hospital, Changde
  - Changsha Central Hospital, Changsha
  - The Second Xiangya Hospital Of Central South University, Changsha
  - The third xiangya hospital of Central South University, Changsha
  - The Third Hospital of Changsha, Changsha
  - Chengdu Second People's Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu
  - Chenzhou No.1 people's Hospital, Chenzhou
  - Affiliated Zhongshan Hospital of Dalian University, Dalian
  - Daqing Oilfield General Hospital, Daqing
  - Daqingshi People's Hospital, Daqing
  - People's Hospital of Deyang City, Deyang
  - The First People's Hospital of Foshan, Foshan
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - No.900 Hospital of PLA Joint Logistics Support Force, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun yet-sen Memorial Hospital, Sun yet-sen Univesity, Guangzhou
  - Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou
  - The Affiliated Panyu Central Hospital of Guangzhou Medical University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Guizhou People's Hospital, Guiyang
  - Hainan General Hospital, Haikou
  - Hangzhou First People's Hospital, Hangzhou
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - Huainan First People's Hospital, Huainan
  - Jiangmen Central Hospital, Jiangmen
  - Center Hospital of Jinan, Jinan
  - Jining No.1 people's hospital, Jining
  - Lanzhou University Second Hospital, Lanzhou
  - Linfen Central Hospital, Linfen
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Luoyang Third People's Hospital, Luoyang
  - Jiangxi Province Integrated Tractional Chinese Medicine& Western Medicine Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanchang People's Hospital, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Nanjing Jiangning Hospital, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Nanyang First People's Hospital, Nanyang
  - Nanyang Second General Hospital, Nanyang
  - Panjin Liao Oil Gem Flower Hospital, Panjin
  - Pingxiang People's Hospital, Pingxiang
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Tongren hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shengyang
  - Shenzhen People's Hospital, Shenzhen
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Union Medical Center Nankai University Affiliated Hospital, Tianjin
  - Wenzhou People's Hospital, Wenzhou
  - Hubei Province Zhongshan Hospital, Wuhan
  - Wuhan Puai Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Shaanxi Provincial People's Hospital, Xi'an
  - Xiangtan Central Hospital, Xiangtan
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - The People's Hospital Of Xuancheng City, Xuancheng
  - The General Hospital of XZCMG (The Second Affiliated Hospital of Xuzhou Medical University), Xuzhou
  - Yanbian University Hospital, Yanji
  - The first People's Hosptal of Yinchuan, Yinchuan
  - Yueyang Central Hospital, Yueyang
  - Yuncheng Central Hospital, Yuncheng
  - The First Affiliated Hospital of Hebei North University, Zhangjiakoou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Colombia (12):
  - Cardiomet CEQUIN S.A.S, Armenia
  - IPS Centro Cientifico-Asistencial S.A.S, Barranquilla
  - Corazon IPS S.A.S., Barranquilla
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - IPS Centro Medico Julián Coronel S.A., Cali
  - Centro De Diagnostico Cardiologico Ltda, Cartagena
  - Fundacion Cardiovascular de Colombia, Floridablanca
  - IPS médicos internistas de Caldas S.A.S., Manizales
  - Fundacion Centro de Investigacion Clinica CIC, Medellín
  - Cardiomet Pereira, Pereira
  - T Y C Inversiones S.A.S Grupsalud, Santa Marta
  - Healthy Medical Center S.A.S, Zipaquirá, Zipaquirá
- Czechia (24):
  - MUDr. Hana Burianova, Bílovec
  - Medicus Services Ltd., Brandýs nad Labem
  - Interni Ordinace s.r.o., Brandýs nad Labem
  - MUDr. Libor Nechvatal s.r.o., Brno
  - St. Anna Hospital, Brno
  - MUDr. Karel Kamenik s.r.o, Brno
  - Vojenska nemocnice Brno, Brno
  - University Hospital Brno, Brno
  - MUDr. Jan Hubac s.r.o., Chrudim
  - Regional Hospital Havlickuv Brod, Havlíčkův Brod
  - Kardiologie KarMa s.r.o, Jablonec nad Nisou
  - Hospital Jihlava, Jihlava
  - MUDr Petra Maskova PhD, Litovel
  - InterKardioML s.r.o., Mariánské Lázně
  - MUDr. Jan Kvasnicka CSc, Prague
  - Kardiologie Vinohrady s r o, Prague
  - Institute for Clinical and Experimental Medicine, Prague
  - University Hospital Motol, Prague
  - University Thomayer´s Hospital, Praha 4-Krc
  - Internist Care s.r.o, Smiřice
  - Kardiologicka ambulance MUDr. Ferkl s.r.o., Trutnov
  - Clinical Trials Services s.r.o, Uherské Hradiště
  - MUDr. Nina Zemkova s.r.o., Uherské Hradiště
  - Cardio Research s.r.o., Zlín
- Germany (26):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Klinikum am Plattenwald, Bad Friedrichshall
  - Studienzentrum Rankestrasse, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Praxis Dr. Toursarkissian, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Vivantes Humboldt-Klinikum, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Praxis Dr. Menzel, Dessau
  - Städtisches Klinikum Dresden, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - ClinPhenomics CVC GmbH, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Praxis Joachim Heisters, Kamp-Lintfort
  - Asklepios Klinik Langen-Seligenstadt GmbH, Langen
  - Praxis Oedeme, Lüneburg
  - Marienhaus Klinikum St. Elisabeth, Neuwied
  - Gemeinschaftspraxis Dres Haggenmiller/Jeserich, Nuremberg
  - Kardiologische Praxis Papenburg, Papenburg
  - Universitätsklinikum Regensburg, Regensburg
  - Praxisgemeinschaft Melcherstätte, Stuhr
  - Gemeinschaftspraxis Dr. Großkopf, Wallerfing
  - Kardiologische Praxis, Wermsdorf, Wermsdorf
- Hungary (22):
  - Lausmed Kft. Outpatient Unit of Internal Medicine, Baja
  - Budai Irgalmasrendi Korhaz, Budapest
  - Obudai Egeszegugyi Centrum Kft., Budapest
  - Belvaros-Lipotvaros Egeszsegugyi Szolgalat, Budapest
  - Geomedical Kft., Budapest
  - Semmelweis University, Budapest
  - Gottsegen National Cardiovascular Center, Budapest
  - Privat Doktor Egeszseguegyi Szolgaltato Zrt., Budapest
  - UNO Medical Trials Kft., Budapest
  - Bekes Varmegyei Koezponti Korhaz, Gyula
  - BKS Research Ltd, Hatvan
  - KomplexLabor Kft., Kecskemét
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - IPR Hungary Kft., Miskolc
  - Dr. Nagy Laszlo Kardiologiai Maganrendeles, Orosháza
  - Coromed-Smo Kft., Pécs
  - Pécsi Tudományegyetem Klinikai Központ, Pécs
  - Da Vinci Private Clinic, Pécs
  - Ujszeged Egeszsegkozpont Diabetes Centrum, Szeged
  - Tolna County Balassa Janos Hospital, Szekszárd
  - Jasz-Nagykun-Szolnok Megyei Hetenyi G. Korhaz-Rendelointezet, Szolnok
  - Belvarosi Egeszseghaz Kft., Zalaegerszeg
- India (14):
  - Kamalnayan Bajaj Hospital, Aurangabad
  - Narayana Institute of Cardiac Sciences, Bangalore
  - Bangalore Medical college, Bengaluru
  - S.P. Medical College & Associated Group of Hospitals, Bikaner
  - Tamil Nadu Government Multi Super Speciality Hospital TNGMSSH, Chennai
  - Apollo Main Hospital, Chennai
  - GNRC Hospital, Guwahati
  - Medanta-The Medicity, Gūrgaon
  - Lisie Hospital, Kochi
  - IPGMER and SSKM Hospital, Kolkata
  - Chopda Medicare and Research Centre Pvt Ltd, Nashik
  - Max Super Speciality Hospital, New Delhi
  - Unicare Heart Institute, Surat
  - King George Hospital, Visakhapatnam
- Italy (8):
  - Humanitas Gavazzeni, Bergamo
  - ASST Papa Giovanni XXIII, Bergamo
  - Az.Osp. Universitaria "Ospedali Riuniti", Foggia
  - Azienda Ospedaliera San Martino, Genova
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - Istituto Clinico Humanitas, Rozzano
- Japan (44):
  - Kasugai Municipal Hospital, Aichi, Kasugai
  - Azumino Red Cross Hospital, Azumino-shi
  - Chiba Heart Clinic, Chiba, Chiba
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Kokura Memorial Hospital, Fukuoka, Kitakyushu
  - National Hospital Organization Hamada Medical Center, Hamada-shi
  - NHO Mito Medical Center, Higashiibaraki-gun
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji-shi
  - Matsuda Cardiovascular Clinic, Hokkaido, Sapporo
  - Oji General Hospital, Hokkaido, Tomakomai
  - Hyogo Prefectural Amagasaki General Medical Center, Hyogo, Amagasaki
  - National Hospital Organization Kanazawa Medical Center, Ishikawa, Kanazawa
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni-shi
  - Kagawa Prefectural Central Hospital, Kagawa, Takamatsu
  - Tokushukai Shonan Kamakura General Hospital, Kamakura-shi
  - Tokushukai Hayama Heart Center, Kanagawa, Miura-gun
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Yokohama Sakae Kyosai Hospital, Kanagawa, Yokohama
  - Mitoyo General Hospital, Kanonji-shi
  - Tokushukai Kishiwada Tokushukai Hospital, Kishiwada-shi
  - North Alps Medical Center Azumi Hospital, Kitaazumi-gun
  - National Hospital Organization Kobe Medical Center, Kobe
  - Shinshu University Hospital, Matsumoto-shi
  - Ehime Prefectural Central Hospital, Matsuyama
  - Matsuyama Shimin Hospital, Matsuyama
  - Mito Saiseikai General Hospital, Mito
  - Hokushin General Hospital, Nakano-shi
  - Okayama City General Medical Center Okayama City Hospital, Okayama, Okayama
  - Naha City Hospital, Okinawa, Naha
  - Urasoe General Hospital, Okinawa, Urasoe
  - Kitano Hospital, Osaka, Osaka
  - Osaka Keisatsu Hospital, Osaka, Osaka
  - Nippon Life Hospital, Osaka, Osaka
  - Japan Community Health care Organization Osaka Hospital, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - NHO Oita Medical Center, Ōita
  - Saga-Ken Medical Centre Koseikan, Saga
  - Sainokuni Higashiomiya Medical Center, Saitama-shi
  - San-Ai Hospital, Saitama-shi
  - NHO Sendai Medical Center, Sendai
  - The University of Osaka Hospital, Suita-shi
  - Tokushima Prefectural Central Hospital, Tokushima
  - Ome Municipal General Hospital, Tokyo, Ome
  - Tomakomai City Hospital, Tomakomai-shi
- Mexico (12):
  - Fundación Cardiovascular de Aguascalientes A.C, Aguascalientes
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Centro Medico Culiacán, Culiacán
  - Centro de Investigacion Biomedica y Farmaceutica, S.C., Distrito Federal
  - CICEJ Centro de Investigacion Clinica Endocrinologica de Jalisco S.C., Guadalajara
  - Salud Cardiovascular, Guadalajara
  - Proactive CR Mexico S.A. de C.V., Irapuato
  - Clinstile S.A. de C.V., México
  - Cardiolink Clin Trials S.C., Monterrey
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Clinical Research Institute S.C., Tlalnepantla
  - Centro de Investigacion Medica Alberto Bazzoni S.A. de C.V., Torreón
- Netherlands (10):
  - Jeroen Bosch Ziekenhuis-Hertogenbosch, 's-Hertogenbosch
  - Rijnstate Hospital, Arnhem
  - Amphia Ziekenhuis, Breda
  - Deventer Ziekenhuis, Deventer
  - Catharina Ziekenhuis, Eindhoven
  - Groene Hart ziekenhuis, Gouda
  - Alrijne Leiderdorp, Leiderdorp
  - St. Antonius Ziekenhuis, Nieuwegein
  - Ikazia Ziekenhuis, Rotterdam
  - De Heel - Zaans Medisch Centrum, Zaandam
- Poland (33):
  - Univ. Clinic Hosp, Bialystok, Bialystok
  - Centrum Medyczne Intercor Sp. z o.o., Bydgoszcz
  - NZOZ Medical Center KERmed, Bydgoszcz
  - Poradnia Kardiologiczna Jaroslaw Jurowiecki, Gdansk
  - Individual Specialist Medical Practice Krzysztof Cymerman, Gdynia
  - Pratia Katowice Medical Center, Katowice
  - Clinical Medical Research Sp. z o.o., Katowice
  - Specialistic Cardiology&Hypertension Out-patient Clin,Kielce, Kielce
  - Leszek Bryniarski Specialized Medical Cabinet, Krakow
  - Linden Sp. z o.o. sp.k., Krakow
  - Beata Miklaszewicz & Dariusz Dabrowski Cardiamed Sp. j., Legnica
  - SANTA FAMILIA Centrum Badan, Profilaktyki i Leczenia, Lodz
  - Individual Specialized Practice, Lodz
  - Lowickie Cardiology Center, Lowicz
  - Velocity Nova Sp. z o.o., Lublin
  - Zanamed Medical Clinic Sp. z o.o., Lublin
  - Medeusz-Plus, Olsztyn
  - Medicome Sp. z o.o., Oświęcim
  - Nzoz Heureka, Piaseczno
  - Non-Public Outpatient Clinic Neuro-Kard Ilkowski & Partners, Poznan
  - Aka-Med Centrum Sp. z o.o. S.K., Ruda Śląska
  - Centrum Medyczne Medyk, Rzeszów
  - Lukmed Lukasz Wozniak, Siedlce
  - Velocity Skierniewice Sp. z o.o, Skierniewice
  - RCMed- Regionalne Centrum Medyczne, Sochaczew
  - NZOZ Procordis, Cardiology Research Center of Sopot, Sopot
  - Velocity Staszow, Staszów
  - FutureMeds Sp. z o.o., Warsaw
  - Balsammedica Sp. z o. o., Warsaw
  - 4. Military Clinical Hospital with Polyclinic SP ZOZ, Wroclaw
  - Sedimed Sp. z o.o., Wroclaw
  - KO-MED Clinical Centers Zamosc, Zamość
  - Centrum Medyczne Serafin med, Żarów
- Romania (16):
  - Spitalul Judetean De Urgenta Dr. Constantin Opris Baia Mare, Baia Mare
  - Spitalul Clinic De Urgenta Prof Dr Agrippa Ionescu, Baloteşti
  - S.C.Centrul Medical Unirea SRL, Brasov
  - Spitalul Judetean de Urgenta Braila, Brăila
  - Emergency University Hospital, Bucharest
  - Clinica Medicala Data Plus SRL, Bucharest
  - S.C. Policlinica CCBR S.R.L., Bucharesti
  - Spitalul Angiocare SRL, Cluj-Napoca
  - Emergency County Hospital Craiova, Craiova
  - S.C.Centrul Medical Unirea S.R.L., Iași
  - Spitalul Clinic Judetean de Urgenta Bihor, Oradea
  - Sal Med Srl, Piteşti
  - Country Clinical Emergency Hospital, Targu-Mures, Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
  - Podoleanu G. Cristian-Gheorghe-Calin, Târgu Mureş
  - S.C Medicali's S.R.L, Timișoara
- Saudi Arabia (5):
  - King AbdulAziz University Hospital, Jeddah
  - King Faisal Specialist Hospital and Research Center, Riyadh
  - King Abdulaziz Medical City, Riyadh
  - King Fahad Medical City, Riyadh
  - King Saud Medical City, Riyadh
- Serbia (11):
  - Clinical Center " Dr Dragisa Misovic Dedinje", Belgrade
  - Clinical Hospital Center Dr. Dragisa Misovic, Belgrade
  - Institute for Cardiovascular diseases Dedinje, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - University Clinical Center of Kragujevac, Kragujevac
  - University Clinical Center Nis, Niš
  - Institute for Treatment and Rehabilitation, Niska Banja, Niška Banja
  - General Hospital Pancevo, Pančevo
  - General Hospital Sveti Luka, Smederevo
  - Health Centre Zajecar, Zaječar
- Slovenia (6):
  - General Hospital Celje, Celje
  - University Hospital Golnik, Golnik
  - General Hospital Jesenice, Jesenice
  - University Medical Center Ljubljana, Ljubljana
  - General Hospital Murska Sobota, Murska Sobota
  - General Hospital Trbovlje, Trbovlje
- South Africa (8):
  - Iatros International, Bloemfontein
  - Josha Research Centre, Bloemfontein
  - TREAD Research, Cape Town
  - Badenhorst, JCW, Centurion
  - Johese Clinical Research: Unitas, Centurion
  - Chris Hani Baragwanath Hospital: Cardiology Department, Johannesburg
  - Dr JM Engelbrecht, Somerset West
  - Clinical Projects Research, Worcester
- South Korea (12):
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wonju-si, Gangwon State
- Spain (12):
  - Hospital Quiron. I.C.U., Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Virgen del Camino, Sanlúcar de Barrameda
  - Complexo Hospitalario Universitario De Santiago, Santiago de Compostela
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Virgen de las Montañas, Villamartin, Cardiz
- Taiwan (10):
  - E-Da Hospital, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Turkey (Türkiye) (14):
  - Çukurova Ü. Tip Fak., Balcali Hastanesi, Kardiyoloji, Adana
  - Afyon Kocatepe University Medical Faculty, Afyonkarahisar
  - Etlik City Hospital, Ankara
  - Firat University Hospital, Elâzığ
  - Ataturk Universitesi Tip Fakultesi, Erzurum
  - Osmangazi Uni Medical Faculty, Eskişehir
  - Gaziantep University Medical Faculty Sahinbey Educational Research Hospital, Gaziantep
  - Siyami Ersek Gogus Kalp ve Damar Cerrahisi Hastanesi, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Medical Park Pendik Hospital, Istanbul
  - Kutahya Health Science University, Kütahya
  - Inonu Universitesi Tip Fakultesi Gogus Hastaliklari ABD, Malatya
  - Mersin University Medical Faculty, Mersin
  - KTU Tip Fakultesi Farabi Hastanesi, Trabzon
- United Kingdom (10):
  - Barnet Hospital, Barnet
  - Southmead Hospital, Bristol
  - Royal Devon and Exeter Hospital, Wonford, Exeter
  - Calderdale Royal Hospital, Halifax
  - Wycombe Hospital, High Wycombe
  - St Bartholomew's Hospital, London
  - The Royal Oldham Hospital, Oldham
  - Northern General Hospital, Sheffield
  - Royal Cornwall Hospital, Truro
  - York and Scarborough Teaching Hospitals NHS Foundation Trust York Hospital, York
- Vietnam (7):
  - Da Nang Hospital, Da Nang
  - Bach Mai hospital, Hanoi
  - Cho Ray Hospital, Ho Chi Minh City
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City
  - Tam Duc Heart Hospital, Ho Chi Minh City
  - Thong Nhat Hospital HCMC, Ho Chi Minh City
  - University Medical Center HCMC, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency